CLINICAL TRIAL: NCT02290158
Title: Effects of a Finishing Protocol Implementation on the American Board of Orthodontics - Objective Grading System Score in Patients of Orthodontic Postgraduate Program: A Quasiexperimental Clinical Trial
Brief Title: Effects of a Finishing Protocol Implementation in Orthodontic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Antioquia (Other)
Responsible Party: Principal Investigator, Alvaro Carvajal, Asociated Pofessor, Universidad de Antioquia
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: BACAZA1
Record Dates: First submitted 2014-10-26; First posted 2014-11-13 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2014-11

CONDITIONS: Malocclusion
Keywords: treatment outcomes; Malocclusion/therapy
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Orthodontic finishing (Active Comparator): Patients receiving a complete orthodontic finishing protocol according to the ABO-OGS
  Interventions: Other: Finishing Protocol
- No orthodontic finishing (No Intervention): Patients receiving orthodontic treatment without the finishing protocol according to the ABO-OGS

INTERVENTIONS:
Other: Finishing Protocol — Students education, cast models and Panoramic X-ray assessment, brackets reposition and frequent clinical evaluation.
  Arms: Orthodontic finishing

SUMMARY:
This study evaluates the effects of a finishing protocol in orthodontic outcomes using ABO-OGS scores. Patients who finish orthodontic treatment and fulfill the inclusion and exclusion criteria receive a treatment using a finishing protocol and their scores are compare with 40 patients who don't receive a finishing protocol

DETAILED DESCRIPTION:
The phase of finishing is the most demanding and detailed of all phases of the orthodontic treatment. American Board of Orthodontics- Objective Grading system is a detailed and objective method that evaluates the quality of the final outcome of orthodontic treatment. In order to evaluate and compare the effects of a protocol implementation on the ABO-OGS scores, standardize cast models and Pan X-Ray from by convenience patients of Orthodontic Postgraduate Program of University of Antioquia who finish orthodontic treatment and receive the protocol are digitized, eight variables are evaluate and ABO-OGS score is calculate. A comparison with 40 no-protocol ABO-OGS scores by convenience-selected patients is done. The protocol includes an educate residents program about finishing problems , an standardized clinical and X-ray assessment , brackets reposition and frequent clinical evaluation. The percentage of the protocol implementation is calculate in every patient and reliability test is make . The descriptive analysis and the ABO-OGS score comparison is done by Pearson or Spearman correlation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who finish orthodontic treatment by orthodontic criteria
* Receive finishing protocol
* Accept and sign inform consent
* Records ( Panoramic Xray and cast models) taken immediately or 7 days after orthodontic appliances are remove

Exclusion Criteria:

* Patients who don't accept being at the study
* Bad quality records
* Prosthodontic, periodontic and surgical needs treatment after orthodontic treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-06; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
ABO-OGS Total Score | Until 7 days after orthodontic appliances are removed
  Sum of 8 variables scores ( alignment, marginal ridge height, buccolingual inclination, overjet, interproximal contact, occlusal contacts, occlusal relationships, and root angulation ) 1: difference less than 1 mm, 2: difference between 1 and 2 mm, 3: difference bigger than 2 mm . Total score less than 20: Excellent , Total score between 20-30: Acceptable and Total Score: > 30 No acceptable

SECONDARY OUTCOMES:
Line Smile | Until 7 days after orthodontic appliances are removed
  Gingival exposure in smiling photo: High: More than 2 mm of gingival exposure, Media: between 2 and O mm of gingival exposure , Low: Less than clinical crown
Arch Smile | Until 7 days after orthodontic appliances are re
  Relationship between incisor borders and upper lower lip border in an smiling photo

CONTACTS AND LOCATIONS:
Locations (1):
- Uniersidad de Antioquia, Medellín, Antioquia, Colombia